CLINICAL TRIAL: NCT00380783
Title: Safety and Efficacy of AGN 203818 for Pain Associated With Painful Bladder Syndrome/Interstitial Cystitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203818-005
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Cystitis, Interstitial
MeSH Terms: conditions — Cystitis, Interstitial

INTERVENTIONS:
Drug: AGN 203818

SUMMARY:
This study will explore the safety and effectiveness of different doses of AGN 203818 in treating the pain associated with painful bladder syndrome/interstitial cystitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of painful bladder syndrome/interstitial cystitis
* Moderate or severe bladder pain

Exclusion Criteria:

* Any other uncontrolled disease
* Pregnant or nursing females

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Reduction in daily pain scores

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma City, Oklahoma, United States